CLINICAL TRIAL: NCT04995835
Title: Ex Vivo Sequestration and Pharmacokinetics of Cefiderocol in Critically Ill Patients Receiving Extracorporeal Membrane Oxygenation (ECMO)
Brief Title: Cefiderocol PK in Patients on ECMO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Joseph L. Kuti, PharmD (Other)
Collaborators: Shionogi Inc. (Industry)
Responsible Party: Sponsor-Investigator, Joseph L. Kuti, PharmD, Director, Center for Anti-Infective Research and Development, Hartford Hospital
Organization: Hartford Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HHC-2021-0086
Record Dates: First submitted 2021-07-30; First posted 2021-08-09 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Sepsis
Keywords: pharmacokinetics; Cephalosporins
MeSH Terms: conditions — Sepsis | interventions — Cefiderocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cefiderocol (Experimental): Participants will receive four to six doses of Cefiderocol as per current prescribing information based on calculated creatinine clearance.
  Interventions: Drug: Cefiderocol

INTERVENTIONS:
Drug: Cefiderocol — After receipt of Cefiderocol, blood samples will be collected at various time points to determine the pharmacokinetics of Cefiderocol
  Other Names: Fetroja

SUMMARY:
Extracorporeal membrane oxygenation (ECMO) is a form of cardiopulmonary life-support for critically ill patients where blood is extracted from the vascular system and circulated by a mechanical pump while it is oxygenated and reinfused into the patient's circulation. It is well known that critically ill patients may experience alterations in antibiotic pharmacokinetics, and as a result, dosing modifications are generally required. There is a need to understand how ECMO circuits affect the pharmacokinetics and disposition of drugs. This study is designed to assess the pharmacokinetics of the new broad-spectrum antibiotic, Cefiderocol, in critically ill patient receiving ECMO.

DETAILED DESCRIPTION:
This is a prospective, open-label, Phase 1b, pharmacokinetic study of Cefiderocol in 8 critically ill patients receiving ECMO support at Hartford Hospital. Informed consent will be collected from all study participants, legal authorized representative, or their next of kin in order to participate. This is not a treatment study; all participants will receive other antibiotics as necessary to treat any current infection.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* On support with veno-venous- or veno-arterial-ECMO

Exclusion Criteria:

* Females who are pregnant or breast-feeding
* History of any moderate or severe hypersensitivity or allergic reaction to any β-lactam antibiotic (a history of mild rash to a cephalosporin followed by uneventful re-exposure is not a contraindication)
* Receiving Cefiderocol to treat documented or suspected infection within 72 hours of screening, or expected to receive Cefiderocol during the study intervention phase
* Severe renal dysfunction defined as a CrCL < 15 mL/min (as calculated by the Cockcroft Gault equation using actual body weight) or requirement for continuous renal replacement therapy or hemodialysis
* A hemoglobin less than 7.2 gm/dl at baseline
* Acute liver injury, defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 5 times the upper limit of normal, or AST or ALT > 3 times the upper limit of normal with an associated total bilirubin > 2 times upper limit of normal
* Any rapidly progressing disease or immediately life-threatening illness (defined as imminent death within 48 hours in the opinion of the investigator)
* Any condition or circumstance that, in the opinion of the investigator, would compromise the safety of the patient or the quality of study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-07-16 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Cefiderocol Clearance | 8 hours
  The Clearance in liters/hour of Cefiderocol from the plasma of critically ill patients receiving ECMO.

SECONDARY OUTCOMES:
Cefiderocol Area Under the Curve (AUC) | 8 hours
  The AUC in milligram*hour/liter of Cefiderocol calculated from concentrations collected between zero and 8 hours at steady-state.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph L Kuti, PharmD, Principal Investigator — Hartford Hospital
Locations (2):
- United States (2):
  - Hartford Hospital, Hartford, Connecticut
  - Columbia University/New York Presbyterian Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: No